CLINICAL TRIAL: NCT02257034
Title: The Effect of Tai Chi in Treating Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chengdu PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yang Min, Ph.D, Chengdu PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TC20140601
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Taichi (Experimental): patients exercise with Tai chi
  Interventions: Other: Taichi
- Control (Sham Comparator): patients under exercise of dance
  Interventions: Other: Dance

INTERVENTIONS:
Other: Taichi
  Arms: Taichi
Other: Dance
  Arms: Control

SUMMARY:
To evaluate the effect of Tai chi on Fibromyalgia

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or older
* meeting the classification of FM per the 1990 ACR criteria
* approval by a healthcare provider for participation

Exclusion Criteria:

* had practiced Tai chi within the past 6 months
* had exercised >30 min three times weekly for past 3 months
* could not independently ambulate without assistive devices
* had BPI pain severity or interference scores less than 5
* had planned elective surgery during study period
* were actively involved in health-related litigation
* were unwilling to keep all treatments/medications steady throughout the study period

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-08; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | up to 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Chengdu Military Area Command PLA, Chengdu, Sichuan, China